CLINICAL TRIAL: NCT07062406
Title: Enhancing Diabetes Care: Implementing Cognitive Behavioral Therapy for Insomnia to Improve Sleep and Cardiometabolic Outcomes
Brief Title: Enhancing Diabetes Care by Treating Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-138
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Type 2; Insomnia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Other: Usual care for diabetes management; Other: Usual care for treatment of insomnia
- Usual Care (Active Comparator)
  Interventions: Other: Usual care for diabetes management; Other: Usual care for treatment of insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — 8 weekly sessions delivered by federally qualified health center behavioral health provider focusing on stimulus control, sleep restriction, and cognitive therapy
  Arms: Cognitive Behavioral Therapy for Insomnia
Other: Usual care for diabetes management — Usual clinical care for management of diabetes (may include pharmacological and non-pharmacological approaches as determined by provider and patient)
Other: Usual care for treatment of insomnia — Usual clinical care for treatment of insomnia (may include pharmacological and non-pharmacological approaches as determined by provider and patient)

SUMMARY:
Insomnia is highly prevalent in individuals with type 2 diabetes (T2D) and is associated with poor glycemic control. Louisiana has one of the highest diabetes prevalence rates in the U.S., with significant disparities by race, income, and rural residence. Despite growing recognition of sleep's role in diabetes management, sleep disturbances remain largely unaddressed in diabetes care. Cognitive behavioral therapy for insomnia (CBT-I) is the first-line treatment for chronic insomnia, yet it is underutilized in primary care clinics such as federally qualified health centers (FQHCs) that serve high-risk populations.

The long-term goal of this research is to improve cardiometabolic health and reduce diabetes disparities by integrating sleep interventions into diabetes care. This pilot study aims to: (1) evaluate the impact of CBT-I on sleep and diabetes-related outcomes, and (2) assess the acceptability, feasibility, and fidelity of implementing an 8-week CBT-I program in an FQHC setting.

The investigators will conduct a randomized controlled trial (RCT) with 30 FQHC patients (aged 40+) with uncontrolled T2D (HbA1c >7%) and comorbid insomnia (Insomnia Severity Index (ISI) score ≥15). Participants will be randomly assigned to either the CBT-I intervention or usual care. Sleep (ISI scores, actigraphy) and cardiometabolic (HbA1c, fasting glucose, insulin) outcomes will be assessed at baseline and three months post-randomization. Implementation success will be evaluated using fidelity, feasibility, and acceptability measures. Findings will provide preliminary evidence for integrating CBT-I into primary care, informing larger trials to improve diabetes outcomes and reduce disparities in Louisiana.

ELIGIBILITY:
Inclusion Criteria:

* aged 40 or older
* receive primary care from participating clinic
* diagnosis of type 2 diabetes
* most recent hemoglobin A1c (HbA1c) >7% within the past year
* Insomnia Severity Index (ISI) score ≥15
* able to speak English

Exclusion Criteria:

* diagnosed or self-reported sleep apnea
* pregnant or planning to become pregnant during the study period
* having a psychiatric or medical condition that would interfere with the ability to complete study procedures
* participating in another diabetes clinical trial
* living in same household as another participant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in change in HbA1c from baseline to 3 months | 3 months
  Difference between intervention and usual care groups in change in hemoglobin A1c (HbA1c) from baseline to 3 months

SECONDARY OUTCOMES:
Between-group difference in change in insomnia symptoms from baseline to 3 months | 3 months
  Difference between intervention and usual care groups in change in Insomnia Severity Index (ISI) score from baseline to 3 months. The ISI is a 7-item questionnaire with scale score ranging from 0 to 28, with higher scores indicating more insomnia symptoms.
Between-group difference in change in fasting glucose from baseline to 3 months | 3 months
  Difference between intervention and usual care groups in change in fasting glucose from baseline to 3 months
Between-group difference in change in concentration of insulin from baseline to 3 months | 3 months
  Difference between intervention and usual care groups in change in concentration of insulin from baseline to 3 months
Between-group difference in change in sleep efficiency from baseline to 3 months | 3 months
  Difference between intervention and usual care groups in change in sleep efficiency from baseline to 3 months. Sleep efficiency will be calculated from wearable device data as the percent of time in bed spent asleep.
Between-group difference in change in wake after sleep onset (WASO) from baseline to 3 months | 3 months
  Difference between intervention and usual care groups in change in wake after sleep onset (WASO) from baseline to 3 months. WASO will be calculated from wearable device data as the number of minutes spent awake after first sleep onset.
Between-group difference in proportion without clinical insomnia symptoms at 3 months | 3 months
  Difference between intervention and usual care groups in proportion with Insomnia Severity Index (ISI) score <15 at 3 months. The ISI is a 7-item questionnaire with scale score ranging from 0 to 28, with higher scores indicating more insomnia symptoms. An ISI score >= 15 indicates symptoms consistent with clinical insomnia.
Between-group difference in change in insomnia symptoms from baseline to 8 weeks | 8 weeks
  Difference between intervention and usual care groups in change in Insomnia Severity Index (ISI) score from baseline to 8 weeks. The ISI is a 7-item questionnaire with scale score ranging from 0 to 28, with higher scores indicating more insomnia symptoms.
Between-group difference in change in sleep efficiency from baseline to 8 weeks | 8 weeks
  Difference between intervention and usual care groups in change in sleep efficiency from baseline to 8 weeks. Sleep efficiency will be calculated from wearable device data as the percent of time in bed spent asleep.
Between-group difference in change in wake after sleep onset (WASO) from baseline to 8 weeks | 8 weeks
  Difference between intervention and usual care groups in change in wake after sleep onset (WASO) from baseline to 8 weeks. WASO will be calculated from wearable device data as the number of minutes spent awake after first sleep onset.
Between-group difference in proportion without clinical insomnia symptoms at 8 weeks | 8 weeks
  Difference between intervention and usual care groups in proportion with Insomnia Severity Index (ISI) score <15 at 8 weeks. The ISI is a 7-item questionnaire with scale score ranging from 0 to 28, with higher scores indicating more insomnia symptoms. An ISI score >= 15 indicates symptoms consistent with clinical insomnia.

CONTACTS AND LOCATIONS:
Locations (1):
- Southeast Community Health Systems, Zachary, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No